CLINICAL TRIAL: NCT05058742
Title: Noninvasive Vagal Nerve Stimulation in Patients With COVID-19 and ARDS for the Reduction of Respiratory, Hemodynamic and Neuropsychiatric Complications
Brief Title: Non-invasive Nervus Vagus Stimulation in Patients With COVID-19 and ARDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Hospital Association (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VNS
Record Dates: First submitted 2021-09-25; First posted 2021-09-28 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: COVID-19; ARDS; Cytokine Storm
Keywords: Nervus vagus stimulation; COVID-19; ARDS; hyperinflammation; cytokine storm
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nervus vagus stimulation (Experimental): Non-invasive Nervus vagus stimulation called AuriStim Intermittent stimluation cycle of three hours of activity and three hours of rest, equating to four cycles of three hours of Stimulation in 24 hours) is performed. The stimulation is performed until the patient's condition is better and he or she isdischarged from OCU or transferred to normal ward or dies.
  Interventions: Device: AuriStim
- Control (No Intervention): There is no Nervus vagus stimulation.

INTERVENTIONS:
Device: AuriStim — Auricular vagal nerve Stimulator, which Targets the auricular branches of the vagal nerve
  Arms: Nervus vagus stimulation

SUMMARY:
Critical ill COVID-19 patients often develop respiratory, hemodynamic and neuropsychiatric complications. An imbalance of sympatho-parasympathetic nervous system is discussed as one of the reasons. The nervus vagus is essential for controlling the sympatho-parasympathetic nervous system and the inflammatory processes.

Aim of this study is to evaluate whether Nervus vagus stimulation decreases the rate of complications (e.g. need of mechanical ventilation, hospital stay, mortality) in critical ill patients.

DETAILED DESCRIPTION:
Introduction:

Critical ill COVID-19 patients often develop respiratory, hemodynamic and neuropsychiatric complications. An imbalance of sympatho-parasympathetic nervous system is discussed as one of the reasons. The nervus vagus is essential for controlling the sympatho-parasympathetic nervous system and the inflammatory processes. A method to stimulate the nervus vagus, is the non-invasive Nervus Vagus Stimulation with AuriStim.

Aims:

Aim of this study is to evaluate whether Nervus vagus stimulation decreases the rate of complications (e.g. need of mechanical ventilation, hospital stay, mortality) in critical ill patients.

Methods:

All patients admitted to ICU at Klinik Favoriten with COVID-19 and moderate to severe ARDS are asked to partcipate. After written consent, a randomisation in Treatment-group (Vagal Nervus Stimulation 4 times a day for each 3 hours until transfer to nomal ward or death) or Non-Treatment-Group is done. In case of stimulation, side effects or intolerance are documented. After discharge or death of the patient, outcomeparameters are evaluated (need of mechanical ventilation, hospital stay, mortality, etc.) and compared between patients of Treatment-Group and Non-Treatment-Group.

ELIGIBILITY:
Inclusion Criteria:

* positive SARS-CoV-2 RT-PCR
* Acute respiratory failure requiring non-invasive respiratory support (NIV or high flow Oxygen)
* PaO2/FiO2 <200

Exclusion Criteria:

* Age <18 years
* Pregnancy (to be excluded using Serum betaHCG in women of childbearing age)
* Signs of infection, eczema or Psoriasis at the application site
* Active malignancy
* Implanted cardiac Pacemaker, deficrillator or other active implanted electrical devices
* Patient unable to consent
* Heart rate <60/min
* Known vagal hypersensitivity
* History of hemophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Nervus vagus stimulation decreases the rate of complications (e.g. need of mechanical ventilation, hospital stay, mortality) | 3 months after admission to ICU
  retrospective analysis after discharge or death or participant

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zoufaly, MD, Principal Investigator — Klinik Favoriten; Eugenijus Kaniusas, Prof. Dr., Study Chair — Vienna University of Technology
Locations (1):
- Klinik Favoriten, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No